CLINICAL TRIAL: NCT04592406
Title: Data on the Prevention of Complications of Prophylactic Intravenous Hydration in Patients With Estimated Glomerular Filtration Rate (eGFR) < 30 ml/Min/1.73m2 From the Maastricht UMC+ Contrast Voorbereidings Polikliniek
Brief Title: Data on the Prevention of Complications of Prophylactic Intravenous Hydration in Patients With eGFR < 30
Acronym: CVP
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL.MUMC.AMACINGrp.4
Record Dates: First submitted 2020-10-07; First posted 2020-10-19 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Acute Kidney Injury (Nontraumatic); Contrast-induced Nephropathy
Keywords: intravascular iodinated contrast administration; prophylactic intravenous hydration
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: CVP screening — An appropriate dual screening process including both renal and cardiac parameters to minimize the risks of post-contrast renal adverse outcomes and of prophylactic hydration in eGFR<30mL/min/1.73m2 patients.

SUMMARY:
At Maastricht University Medical Centre (Maastricht UMC+) a specialised unit was established where a dual screening process including both renal and cardiac parameters is used to minimize the risk of contrast-induced acute kidney injury as well as the risk of prophylactic hydration in eGFR<30mL/min/1.73m2 patients. Very little data exists on patients with eGFR <30mL/min/1.73m2 in this context. The current study aims to describe post-contrast outcomes of patients to whom this screening method has been applied.

DETAILED DESCRIPTION:
A large retrospective observational study, including 4-years of elective procedures with intravascular iodinated contrast administration in eGFR<30mL/min/1.73m2 patients at Maastricht UMC+, found that prophylactic intravenous hydration might confer some benefit for renal function. For patients who had received prophylactic hydration, adjusted odds ratios for risk of post-contrast acute kidney injury, and 1-month eGFR decline and dialysis were all lower than 1. These results were not significant, but suggest that hydration may be protective. On the other hand, adjusted odds ratios for all-cause mortality within 1-month post-contrast were higher than 1, with point estimates indicating a trend toward higher risk of short-term mortality after prophylaxis as compared to no prophylaxis. Confounding by indication may be responsible for the observed increased risk of short-term mortality, but complications of the prophylaxis did contribute towards the risk. Amongst the 281 eGFR<30mL/min/1.73m2 prophylaxis patients studied, 18 (6.4%) serious complications occurred: 3 arrhythmias, and 15 heart failures including 5 deaths. Of all 21 deaths recorded for the prophylaxis patients, 24% (5/21) were considered to be related to intravenous fluids. An exploration of differences in baseline characteristics between patients with and without serious complications suggested that these can be avoided if cardiac function parameters are given extra and individual attention before deciding whether to administer prophylaxis to high-risk patients with eGFR<30mL/min/1.73m2. At Maastricht UMC+ a specialised unit (called the CVP) was established where a dual screening process including both renal and cardiac parameters is used to minimize the risk of contrast-induced acute kidney injury as well as the risk of prophylactic hydration in eGFR<30mL/min/1.73m2 patients. In order to enable real function follow-up, the CVP registers data on all patients with eGFR <30 receiving intravascular iodinated contrast material, including acute patients who did not receive the dual screening process prior to prophylactic intravenous hydration. The current study aims to describe post-contrast outcomes of patients to whom the CVP screening method has been applied and to compare them to earlier outcomes of patients to whom the screening was not applied.

ELIGIBILITY:
Inclusion Criteria:

* eGFR <30 mL/min/1.73m2 in absence of dialysis
* referred for a procedure with intravascular administration of iodinated contrast material at Maastricht UMC+

Exclusion Criteria:

* age <18 years
* dialysis or pre-dialysis
* emergency or intensive care status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with eGFR <30 mL/min/1.73m2 in absence of dialysis referred for a procedure with intravascular administration of iodinated contrast material at Maastricht UMC+
Sampling Method: Non-Probability Sample
Enrollment: 443 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2023-01-06 (Actual); Study Completion 2023-01-06 (Actual)

PRIMARY OUTCOMES:
complications of prophylactic intravenous hydration | 14 days
  serious complications of prophylactic intravenous hydration (heart failure, arrhythmia)
complications of prophylactic intravenous hydration 2 | 14 days
  deaths with primary cause heart failure (and no known other underlying cause) within 14 days post-contrast
complications of prophylactic intravenous hydration 3 | 14 days
  proportion of all deaths in prophylaxis subgroups with primary cause heart failure within 14 days

SECONDARY OUTCOMES:
incidence of post-contrast acute kidney injury | 6 days
  acute increase in serum creatinine within 5 days post-contrast
incidences of 1-month post-contrast dialysis and mortality | 35 days
  incidences of dialysis and all-cause mortality within post-contrast
post-contrast change in eGFR | 6 days
  change in eGFR from baseline post-contrast
prophylaxis administered | 1 day
  percentage of patients receiving standard, adapted and no prophylactic intravenous hydration
post-contrast AKI according to KDIGO definition | 6 days
  post-contrast AKI according to KDIGO definition
ODDS ratios prophylaxis | 1 month
  where possible odds ratios for standard prophylaxis versus no prophylaxis and adapted prophylaxis versus no prophylaxis will be calculated for post-contrast acute kidney injury, 1-month dialysis and death

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht UMC, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No